CLINICAL TRIAL: NCT04215172
Title: Safety and Efficacy of Long-Term Macrolide Therapy in Patients With COPD-Bronchiectasis Overlap Syndrome
Brief Title: Macrolides in COPD- Bronchiectasis Overlap
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Sayed Ali, Assistant Lecturer, Assiut University
Other Study IDs: COPD_bronchiactasis
Record Dates: First submitted 2019-12-18; First posted 2020-01-02 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Macrolides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- macrolides group: Every patient of this group will be educated and instructed about usage, dosing and side effects of the drug.
  Dose: azithromycin 500 mg three times weekly for 6 months. added to the conventional treatment.
  Interventions: Drug: Macrolides
- conventional group: Every patient of this group will receive the conventional treatment.

INTERVENTIONS:
Drug: Macrolides — administration of azithromycin three times weekly for six months
  Groups: macrolides group

SUMMARY:
To assess safety of long-term macrolide therapy in patients with COPD-bronchiectasis overlap syndrome And evaluate its efficacy in treating COPD-bronchiectasis overlap syndrome regarding change in clinical, functional and microbiological profile.

To define the, clinical, radiological, functional and microbiological patterns of patients with COPD-bronchiectasis overlap syndrome

DETAILED DESCRIPTION:
COPD and bronchiectasis share common symptoms of cough with sputum production and susceptibility to recurrent exacerbations driven by new or persistent infection The overlap between chronic obstructive pulmonary disease (COPD) and bronchiectasis is a neglected area of research, and it is not covered by guidelines for clinical practice COPD is diagnosed on the basis of poorly reversible airflow obstruction and is therefore a physiological diagnosis. It is defined when an objective measure of airflow obstruction is associated with an abnormal inflammatory response of the lung to noxious stimuli, with cigarette smoke being the most common exposure in the developed world. Operationally, this implies that patients with any sufficient exposure and fixed airflow obstruction are labelled as having COPD.

Bronchiectasis is diagnosed in the presence of airway dilatation and airway wall thickening on imaging (usually computed tomography (CT)), and is therefore a structural diagnosis. Clinically significant disease is present when imaging abnormalities are associated with symptoms of persistent or recurrent bronchial infection.

in the 2014 Global initiative for chronic Obstructive Lung Disease guidelines, bronchiectasis was for the first time defined as a comorbidity of chronic obstructive pulmonary disease (COPD), and this change has been retained in the 2015 update, which emphasizes the influence of bronchiectasis in the natural history of COPD.

The prevalence of bronchiectasis in patients with COPD is high, especially in advanced stages. The identification of bronchiectasis in COPD has been defined as a different clinical COPD phenotype with greater symptomatic severity, more frequent chronic bronchial infection and exacerbations, and poor prognosis.

A recent meta-analysis by Du et al, of 5,329 COPD patients found a greatly increased exacerbation risk due to comorbid COPD with bronchiectasis compared to COPD alone.18 Moreover, the risk of exacerbations rose almost two times higher, colonization of the lungs four times higher, severe airway obstruction 30 percent higher, and mortality two times higher. It is not surprising that such elevated risks are also associated with higher healthcare costs.

Treatments useful in COPD may not be widely effective in bronchiectasis and vice versa. Inhaled corticosteroids provide perhaps the best example of this: they are widely used in COPD but not recommended for most patients with bronchiectasis . The reasons for this are unclear but probably reflect, in part, the diverse aetiology underlying bronchiectasis. In contrast, inhaled antibiotics, including antipseudomonal agents in appropriate patients, are of benefit and appear in current bronchiectasis guidelines ,but are not used routinely in stable COPD Macrolides, in addition to their antimicrobial effects, have decreased neutrophil chemotaxis and infiltration into the respiratory epithelium, inhibition of transcription factors leading to decreased proinflammatory cytokine production, down-regulation of adhesion molecule expression, inhibition of microbial virulence factors including biofilm formation, reduced generation of oxygen-free radicals, enhanced neutrophil apoptosis, and decreased mucus hypersecretion with improved mucociliary clearance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above, male or female.
* Non / Ex-smokers.
* Confirmed diagnosis of bronchiectasis based on high-resolution computed tomography scan.
* Confirmed diagnosis of COPD based on pulmonary function test.

Exclusion Criteria:

* Active smokers.
* Moderate to severe liver impairment (Child-Pugh B or C) and/or sever renal impairment (c. clearance less than 30ml/min).
* Patients who are known to be hypersensitive to macrolide.
* Patient with known or susceptible to have rhythm problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are admittted toChest department of Assiut University Hospitals or visit its outpatients' clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
long-term macrolides therapy in patients with COPD-bronchiectasis overlap syndrome regarding ototoxicity, hepatotoxicity and cardiac toxicity | two years
  1)-ototoxicity by whispered- voice test before starting treatment and monthly The examiner stands arm's length (0.6 m) behind the seated patient and whispers a combination of numbers and letters (for example, 4-K-2) and then asks the patient to repeat the sequence.
  If the patient responds correctly, hearing is considered normal; if the patient responds incorrectly, the test is repeated using a different number/letter combination The examiner always stands behind the patient to prevent lip reading The other ear is assessed similarly with a different combination of numbers and letters
  -2)-assessment of hepatotoxicity by measuring liver enzymes (aspartate transaminase AST, Alanine transaminase ALT (Unit/Liter)) before starting treatment and monthly.
  3)-assessment of possible prolongation of QT interval (millimeters) by ECG (electrocardiogram) before starting treatment and monthly.
evaluate macrolides in treating COPD-bronchiectasis overlap syndrome regarding improvement of symptoms, frequency of exacerbations, systemic inflammatory response and pulmonary function tests. | two years
  * symptoms:
    1. Dyspnea score by mMRC (modified medical research council) score, with strenuous exercise 0 when hurrying or walking up a slight hill +1 Walks slower than people of the same age because of dyspnea +2 Stops for breath after walking 100 yards +3 Too dyspneic to leave house +4
    2. sputum volume by (milliliter),
    3. bronchiectasis health questionnaire (BHS)
  * exacerbation: Frequency of outpatient visits per month and hospital admission if happened (number\month).
  * systemic inflammation:
    1. CBC (complete blood count) (White Blood Cells(n/ microliter), differential count (%)
    2. Erythrocyte Sedimentation Rate (millimeter/hour)
    3. C-Reactive Protein (milligram\ liter)
  * Microbiological:
  Change in microbiological picture based on sputum culture and sensitivity
  - Functional: Change in FEV1 (forced expiratory volume at one second) (liter/second.) all these will be done before starting treatment and monthly.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hurst JR, Elborn JS, De Soyza A; BRONCH-UK Consortium. COPD-bronchiectasis overlap syndrome. Eur Respir J. 2015 Feb;45(2):310-3. doi: 10.1183/09031936.00170014. No abstract available. PMID 25653262
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Martinez-Garcia MA, Miravitlles M. Bronchiectasis in COPD patients: more than a comorbidity? Int J Chron Obstruct Pulmon Dis. 2017 May 11;12:1401-1411. doi: 10.2147/COPD.S132961. eCollection 2017. PMID 28546748
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Background] Ni Y, Shi G, Yu Y, Hao J, Chen T, Song H. Clinical characteristics of patients with chronic obstructive pulmonary disease with comorbid bronchiectasis: a systemic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2015 Jul 28;10:1465-75. doi: 10.2147/COPD.S83910. eCollection 2015. PMID 26251586
- [Background] Figueiredo Bde C, Ibiapina Cda C. The role of macrolides in noncystic fibrosis bronchiectasis. Pulm Med. 2011;2011:751982. doi: 10.1155/2011/751982. Epub 2011 Sep 5. PMID 22292118
- [Background] Chalmers JD. Bronchiectasis and COPD Overlap: A Case of Mistaken Identity? Chest. 2017 Jun;151(6):1204-1206. doi: 10.1016/j.chest.2016.12.027. No abstract available. PMID 28599926